CLINICAL TRIAL: NCT01562106
Title: A Prospective Investigation of the Use of Fluorescence Imaging on the da Vinci Surgical System for Ultrastaging of Endometrial Cancer by Sentinel Node Assessment
Brief Title: Investigating the Use of Fluorescence Imaging in Endometrial Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IR 5197
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Endometrial Cancer
Keywords: Cancer of Endometrium; Cancer of the Endometrium; Carcinoma of Endometrium; Endometrial Carcinoma; Endometrium Cancer; Neoplasms, Endometrial
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG Dye (Experimental): Fluorescence-guided sentinel lymph node detection
  Interventions: Procedure: Fluorescence-guided sentinel lymph node detection

INTERVENTIONS:
Procedure: Fluorescence-guided sentinel lymph node detection — During standard endometrial cancer surgery, ICG dye will be injected into the cervix to identify sentinel lymph nodes in the pelvis.

SUMMARY:
The main purpose of the study is to evaluate the detection rate and accuracy of fluorescence imaging in endometrial cancer staging by sentinel node assessment.

DETAILED DESCRIPTION:
In many cancer types, such as breast cancer and melanoma, sentinel node assessment has become the standard of care surgical treatment. Sentinel nodes are the first lymph nodes to which cancer cells are likely to spread from a primary tumor. Removal of a sentinel node for examination accurately predicts whether the cancer has spread to other nodes further along in the nodal chain. Fluorescence imaging with ICG dye (Indocyanine Green) has been used to detect lymph nodes in patients with gastric, colorectal and breast cancer. To date, the use of this technique in endometrial cancer has not been reported.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven endometrial carcinoma
* Must have planned to undergo standard endometrial cancer staging surgery as part of their routine clinical care
* Must be 18 years of age and older
* Must be able to comply with all the study procedures

Exclusion Criteria:

* Significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests, with total bilirubin > 1.5 times normal, and/or SGOT > 2 times normal
* Uremia, serum creatinine > 2.0 mg/dl
* Previous history of adverse reaction or allergy to ICG dye, iodine, shellfish, or iodine dyes
* Previous lymphadenectomy or surgery that could change the uterine lymphatic drainage
* Pregnant
* Currently participating in a drug, biologic and/or device treatment study
* Any medical condition that would normally prevent someone from receiving general anesthesia or undergoing standard surgical procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evaluating detection rate and accuracy of fluorescence-guided sentinel lymph node detection in endometrial cancer. | Average expected time of 12 weeks

SECONDARY OUTCOMES:
Determine the rate of upstaging using fluorescence-guided sentinel lymph node assessment by microscopic evaluation. | Average expected time of 12 weeks
  In cancer, "upstaging" is changing the stage used to describe a patient's cancer from a lower stage (less extensive) to a higher stage (more extensive). The sentinel lymph nodes removed during the flourescence guided surgery will be examined microscopically to determine how often upstaging occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Paley, MD, Principal Investigator — Swedish Medical Center
Locations (3):
- United States (3):
  - Swedish Medical Center Issaquah Campus, Issaquah, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington